CLINICAL TRIAL: NCT06736808
Title: Assessment of Patient Understanding of Educational Material at Above and Below a Sixth Grade Reading Level
Brief Title: Patient Understanding of Handouts at Different Reading Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-2684
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Health Literacy
Keywords: readability; patient understanding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Below Sixth Grade Reading Level (Experimental): Participants randomized to this experimental arm will read a simplified handout on pelvic organ prolapse written at below a sixth grade reading level.
  Interventions: Other: Handout Written at Below a Sixth Grade Reading Level
- Above Sixth Grade Reading Level (Active Comparator): Participants randomized to this control arm will read a standard handout on pelvic organ prolapse written at above a sixth grade reading level.
  Interventions: Other: Handout Written at Above a Sixth Grade Reading Level

INTERVENTIONS:
Other: Handout Written at Below a Sixth Grade Reading Level — Participants randomized to this experimental arm will read a simplified handout on pelvic organ prolapse written at below a sixth grade reading level.
  Arms: Below Sixth Grade Reading Level
Other: Handout Written at Above a Sixth Grade Reading Level — Participants randomized to this control arm will read a standard handout on pelvic organ prolapse written at above a sixth grade reading level.
  Arms: Above Sixth Grade Reading Level

SUMMARY:
The goal of this randomized clinical trial is to learn if participants are better able to understand medical handouts written at below a sixth grade reading level compared to those written at above a sixth grade reading level. The main question it aims to answer is:

• Do participants score higher on a knowledge test after reading a handout written at below a sixth grade reading level compared to after reading a handout written at above a sixth grade reading level?

Researchers will compare knowledge scores on pelvic organ prolapse after participants read a handout written at an eight grade reading level compared to the same handout re-written to be at a fifth grade reading level.

Participants will:

* Read a one page handout (written at either above or below a sixth grade reading level) on pelvic organ prolapse
* Complete a one page multiple-choice test on pelvic organ prolapse

DETAILED DESCRIPTION:
The secondary objective is to determine characteristics of patients whose knowledge levels are higher after reading educational material written below a sixth grade reading level compared to material written above a sixth grade reading level.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to complete pen and paper questionnaire

Exclusion Criteria:

* Unable to understand or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Knowledge Assessment Score | Assessed during completion of a 5 minute survey after reading a one page informational handout for approximately 10 minutes
  Mean number of correct answers from 0 to 12 on the validated Prolapse Knowledge Questionnaire where 0 indicates 0 correct answers (worst knowledge score) and 12 indicates all correct answers (best knowledge score).
Participant-reported Handout Utility | Assessed during completion of a 5 minute survey after reading a one page informational handout for approximately 10 minutes
  Percentage of participants who respond "Yes" that reading the handout increased their understanding of pelvic organ prolapse on a Yes/No/Don't know scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bertie Geng, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina Urogynecology and Reconstructive Pelvic Surgery at REX, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 12 months following publication until 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Shah AD, Massagli MP, Kohli N, Rajan SS, Braaten KP, Hoyte L. A reliable, valid instrument to assess patient knowledge about urinary incontinence and pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Sep;19(9):1283-9. doi: 10.1007/s00192-008-0631-x. Epub 2008 May 15. PMID 18480958